CLINICAL TRIAL: NCT04599712
Title: Pre-Approval Access With Amivantamab in Patients With Metastatic Non-Small Cell Lung Cancer With EGFR Exon 20 Insertion Mutations Who Have Failed Platinum-Based Chemotherapy
Brief Title: Pre-Approval Access With Amivantamab (JNJ-61186372) in Participants With Metastatic Non-Small Cell Lung Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108905; 61186372LUC4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — amivantamab

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Amivantamab — Amivantamab will be administered intravenously at the recommended doses based on weight (1050 milligram [mg] or 1400 mg) once weekly for the first 4 week cycle (1 cycle equals to 28 days), then every 2 weeks thereafter.
  Other Names: JNJ-61186372

SUMMARY:
The purpose of this expanded access program (EAP) is to provide amivantamab for the treatment of participants with metastatic non-small cell lung cancer who have epidermal growth factor receptor exon 20 insertion mutations, and whose disease has progressed during or after current standard of care platinum-based chemotherapy. This intermediate EAP may be considered for individuals with serious/life-threatening diseases or conditions, where there are no alternative treatments or where individuals have progressed following standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed unresectable or metastatic non-small cell lung (NSCLC) cancer with an epidermal growth factor receptor (EGFR) exon 20 insertion (Exon20ins), not amenable to curative therapy
* Has completed prior treatment with platinum-based chemotherapy. In the case of platinum ineligible participants, the participant may qualify if previously treated with an alternative treatment (example, an investigational or approved EGFR Exon 20 targeted tyrosine kinase inhibitor [TKI], or see guidelines such as those from national comprehensive cancer network [NCCN] or European society for medical oncology [ESMO] for alternative non-platinum-based treatments)
* Life expectancy is projected to be greater than or equal to (>=) 3 months with adequate hepatic, renal, pulmonary and cardiac function (physician assessed)

Exclusion Criteria:

* Has medical history of interstitial lung disease (ILD), including drug-induced ILD or radiation pneumonitis requiring treatment with prolonged steroids or other immune suppressive agents within the last 3 months
* Has leptomeningeal disease that is active or symptomatic
* Symptomatic, unstable or untreated brain metastases (need to be resolved prior to participating in the program)
* Known allergies, hypersensitivity, or intolerance to amivantamab or its excipients or to other monoclonal antibodies
* Is pregnant or breastfeeding

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC